CLINICAL TRIAL: NCT01516762
Title: Radium-223 Chloride (BAY88-8223) in Castration-Resistant (Hormone-Refractory) Prostate Cancer Patients With Bone Metastases
Brief Title: Radium-223 Dichloride (BAY88-8223) in Castration-Resistant (Hormone-Refractory) Prostate Cancer Patients With Bone Metastases
Status: No longer available | Type: Expanded Access
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15995; 2011-004469-33 (EudraCT Number)
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Prostatic Neoplasms
Keywords: Radium 223; Alpharadin; Prostate Cancer; Bone metastases; Castrate resistant prostate cancer; Hormone refractory prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride

INTERVENTIONS:
Drug: Radium-223 dichloride (BAY88-8223) — One injection to be administered every 4 weeks up to 6 injections. The dose per injection is 50 kBq/kg body weight.

SUMMARY:
This study is a prospective, interventional, open-label, multi-center early access program for the use of Ra-223 Cl2 in HRPC/CRPC patients diagnosed with symptomatic bone metastasis and to collect additional short and long term safety data on the product.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically or cytologically confirmed prostate cancer
* Patients diagnosed with symptomatic progressive bone predominant metastatic CRPC/HRPC with at least 2 skeletal metastases on imaging with no lung, liver, and/or brain metastasis (lymph node only metastasis is allowed)
* Symptomatic is defined as either

  * Regular (not occasional) use of analgesic medication for cancer related bone pain (≥ level 1; World Health Organization [WHO] ladder for cancer pain), or
  * Treatment with external beam radiation therapy (EBRT) for bone pain (the EBRT should be within the last 12 weeks before treatment)
* Progressive disease is defined either by:

  * The appearance of new bone lesions. If progression is based on new lesion(s) on imaging only without an increase in prostate specific antigen (PSA), then PSA values from 3 assessments within the last 6 months must be provided; OR
  * In the absence of new bone lesions, 2 subsequent increases in serum PSA over previous reference value, which should not be more than 6 months before screening, each measured at least 1 week apart with the last PSA ≥ 5 ng/mL. (The reference value time point 1, is defined as the last PSA measured before increases are documented, with subsequent values obtained a minimum of 1 week apart. If the PSA at time point 3 is greater than the PSA at time point 2, then eligibility has been met. If the PSA at time point 3 is not greater than the PSA at time point 2 but, the PSA value at time point 4 and/or time point 5 is greater than the PSA at time point 2, the patient is eligible assuming that other criteria are met).
* No intention to use cytotoxic chemotherapy within the next 6 months
* Life expectancy ≥ 6 months
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2
* Adequate hematological, liver, and renal function

  * Absolute neutrophil count (ANC) ≥ 1.5 x10^9/L
  * Platelet count ≥ 100 x10^9/L
  * Hemoglobin ≥ 10.0 g/dL (100 g/L; 6.2 mmol/L)
  * Total bilirubin level ≤ 1.5 x institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
  * Creatinine ≤ 1.5 x ULN
  * Albumin > 25 g/L *Any bone imaging techniques as per institutional standard of care

Exclusion Criteria:

* Treatment with an investigational drug within previous 4 weeks, or planned during the treatment period or follow-up
* Eligible for first course of docetaxel, i.e., patients who are fit enough, willing, and who are located where treatment with docetaxel is available
* Treatment with cytotoxic chemotherapy within previous 4 weeks prior to screening, or failure to recover from adverse events (AEs) due to cytotoxic chemotherapy administered more than 4 weeks previous prior to screening (however, ongoing neuropathy is permitted)
* Prior hemibody external radiotherapy is excluded. Patients who received other types of prior external radiotherapy are allowed provided that the bone marrow function is assessed and meets the protocol requirements for hemoglobin, absolute neutrophil count, and platelets
* Received systemic therapy with radionuclides (e.g., strontium-89, samarium-153, rhenium-186, or rhenium-188, or radium-223 dichloride) for the treatment of bony metastases
* Other malignancy treated within the last 3 years (except non melanoma skin cancer or low-grade superficial bladder cancer)
* Visceral metastases as assessed by abdominal or pelvic computed tomography (CT) (or other imaging modality based on institutional standard of care)
* Presence of brain metastases
* Lymphadenopathy exceeding 6 cm in short-axis diameter
* Any size pelvic lymphadenopathy if it is thought to be a contributor to concurrent hydronephrosis.
* Imminent spinal cord compression based on clinical findings and/or magnetic resonance imaging (MRI). Patients with history of spinal cord compression should have completely recovered.
* Any other serious illness or medical condition, such as but not limited to:

  * Any infection ≥ National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 Grade 2
  * Cardiac Failure New York Heart Association (NYHA) Class III or IV
  * Crohn's disease or ulcerative colitis
  * Bone marrow dysplasia
* Fecal incontinence

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (51):
- United States (51):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Greenbrae, California
  - La Jolla, California
  - San Francisco, California
  - Stanford, California
  - Aurora, Colorado
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Fort Myers, Florida
  - Miami Beach, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Goshen, Indiana
  - Iowa City, Iowa
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Rockville, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Las Vegas, Nevada
  - New Brunswick, New Jersey
  - Newark, New Jersey
  - New Hyde Park, New York
  - New York, New York
  - Syracuse, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Springfield, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Myrtle Beach, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Hampton, Virginia
  - Norfolk, Virginia
  - Seattle, Washington
  - Wheeling, West Virginia
  - Milwaukee, Wisconsin